CLINICAL TRIAL: NCT01617772
Title: Comparison the Effectiveness of L-Carnitine With Atorvastatin in Non-Alcoholic Steatohepatitis (NASH)
Brief Title: Atorvastatin, L-Carnitine and Non-Alcoholic Steatohepatitis
Acronym: NALCAT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 90-03-37-15428
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: Non-alcoholic steatohepatitis, Atorvastatin, L-Carnitine
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Atorvastatin; Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Atorvastatin (Experimental): 20mg atorvastatin daily
  Interventions: Drug: Atorvastatin
- Carnitine (Experimental): 1000mg L-carnitine daily
  Interventions: Drug: L-Carnitine
- Atoral (Experimental): 1000mg L-carnitine and 20mg atorvastatin
  Interventions: Drug: Atorvastatin; Drug: L-Carnitine
- Placebo (Placebo Comparator): Identically looking placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 20 mg
  Arms: Atoral; Atorvastatin
Drug: L-Carnitine — 1000mg L-carnitine
  Arms: Atoral; Carnitine
Drug: Placebo — Identically looking placebo
  Arms: Placebo

SUMMARY:
The aim of the present study was to compare the effects of simvastatin and L-carnitine coadministration versus simvastatin, L-Carnitine monotherapy on liver transaminases and liver elasticity in NASH patients.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) represents a spectrum of disease ranging from steatosis to steatohepatitis (nonalcoholic steatohepatitis, NASH) to cirrhosis. Statins are competitive inhibitors of Hydroxymethylglutaryl-CoA reductase, the rate-limiting step in cholesterol biosynthesis. They occupy a portion of the binding site of Hydroxymethylglutaryl-CoA, blocking access of this substrate to the active site on the enzyme. A reduction in intrahepatic cholesterol leads to an increase in LDL receptor turnover that results from an enhanced rate of hepatic LDL receptor cycling. On the other hand recent studies have implicated several important cellular processes and signaling pathways that are affected by abnormal lipid metabolism, resulting in specific biochemical, histological, and clinical changes associated with NAFLD.

Maybe statins, as lipid lowering agents, and through their effect in reduction of intrahepatic cholesterol, can affect the abnormal lipid metabolism in NASH.

L- carnitine, can improve the outcome of NASH, because it reduces lipid levels, limits oxidative stress, and modulates inflammatory responses . It performs a number of essential intracellular and metabolic functions, such as fatty acid transport, detoxification of potentially toxic metabolites, regulation of the mitochondrial acyl-CoA / CoA ratio, and stabilization of cell membranes. It has a pivotal role in the transport of long chain fatty acids across the inner mitochondrial membrane.

ELIGIBILITY:
Inclusion Criteria:

* NASH diagnosed on the basis of the following criteria:

  1. Imaging techniques showing evidence of hepatic steatosis
  2. Increased alanine transaminase above 1.5 times normal (normal: 20 IU/L for women, 30 for men) on two occasions three months apart.

Exclusion Criteria:

* Patients with hepatitis B or C
* alanine transaminase > 300 IU/L
* Participants presenting one or more causes commonly associated with secondary NAFLD (drugs, surgical procedures, environmental toxins, or total parenteral nutrition)
* Alcohol ingestion greater than 40 gr per week
* Abnormal Lipid profile (TG>500 , LDL>160)
* Patients with hypertension, diabetes mellitus, coronary heart disease
* Fibroscan score more than 14 kp
* pregnancy, lactation
* Drug addiction
* Reynolds Risk Score > 10%
* Not consenting to the study

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
improvement in liver stiffness | 2 years
  As measured by Fibroscan

SECONDARY OUTCOMES:
improvement in liver enzyme levels | 2 years
  Difference between last and first measurements
Adverse drug events | 2 years
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, MD, Study Chair — Tehran University of Medical Sciences
Locations (2):
- Iran (2):
  - Pars Cohort Center, Shiraz, Fars
  - Masoud Clinic, Tehran